CLINICAL TRIAL: NCT00342147
Title: Family Study of Head and Neck Cancers in Taiwan
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995046; OH95-C-N046
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Nasopharyngeal Neoplasms; Herpesvirus 4, Human
Keywords: EBV; NPC
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected: blood and saliva.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: This is a high risk population of families for NPC

SUMMARY:
Nasopharyngeal carcinoma is a rare tumor among Caucasians which occurs with high incidence among individuals of Chinese descent. The disease is believed to have a multifactorial etiology with genetic, viral, and other environmental factors being involved. Little is known, however, about the genetic component of this disease.

We have recently completed subject recruitment for a case-control study of NPC in Taiwan. Using information obtained from the NPC cases recruited into this NCI-sponsored case-control study as well as from a parallel cross-sectional study conducted by our Taiwanese collaborators, we have been able to identify 120-150 families with multiple family members affected with NPC.

The purpose of the study described herein is to determine the role of inherited genetic factors in the etiology of NPC and to examine the effect of these genetic susceptibility factors on risk associated with environmental exposures.

Families will initially be contacted via the proband who previously participated in our case-control and cross-sectional studies. Subsequently, informative family members will be asked to visit the study clinic to participate in the study. A family history questionnaire will be administered to the proband from each of the families selected for study. In addition, a risk factor questionnaire will be administered to all participating family members, and 30-40 ml of blood and an oral sample will be obtained from each study participant. Additional study components include medical record review to verify the diagnosis of NPC, retrieval of tumor tissue blocks as a source of DNA for study, and clinical exams on a sample of unaffected individuals to exclude the possibility of prevalent, undetected disease among family members.

Oral and laryngeal cancer families will also be recruited in a manner similar to that described for NPC families, in an attempt to elucidate genetic factors linked to the development of these two cancers....

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma is a rare tumor among Caucasians that occurs with high incidence among individuals of Chinese descent. The disease is believed to have a multifactorial etiology with genetic, viral, and other environmental factors being involved. Little is known, however, about the genetic component of this disease.

We previously completed a case-control study of NPC in Taiwan. Using information obtained from the NPC cases recruited into this NCI-sponsored case-control study and parallel sources, we have been able to identify 250 families with multiple family members affected with NPC.

The purpose of the study described herein is to determine the role of inherited genetic factors in the etiology of NPC and to examine the effect of these genetic susceptibility factors on risk associated with environmental exposures.

Families will initially be contacted via an affected proband. Subsequently, informative family members will be asked to visit the study clinic to participate in the study. A family history questionnaire will be administered to the proband and other affected family members from each of the families selected for study. In addition, a risk factor questionnaire will be administered to all participating family members, and 30-40 ml of blood and an oral sample will be obtained from each study participant. Additional study components include medical record review to verify the diagnosis of NPC, retrieval of tumor tissue blocks as a source of DNA for study, and clinical exams on a sample of unaffected individuals to exclude the possibility of prevalent, undetected disease among family members.

Oral and laryngeal cancer families will also be recruited in a manner similar to that described for NPC families, in an attempt to elucidate genetic factors linked to the development of these two cancers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects with head and neck cancer who are participants in the case-control study of NPC or the parallel studies of head and neck cancers conducted by the Taiwanese.

Subjects who report one or more first degree family members affected with NPC, oral cancer, or laryngeal cancer.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a high risk population of families for NPC
Sampling Method: Non-Probability Sample
Enrollment: 3795 (Actual)
Dates: Start 1995-11-07 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
Nasopharyngeal Carcinoma | Ongoing
  Nasopharyngeal carcinoma diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Allan Hildesheim, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Taiwan University College of Medicine, Taipei, Taiwan, China